CLINICAL TRIAL: NCT06741644
Title: A Phase I/II, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activities of CS2009, a Tri-specific Antibody Targeting PD-1/VEGFA/CTLA-4, as Monotherapy and Combination Therapy in Participants With Advanced Solid Tumors
Brief Title: A Phase I/II Study of CS2009 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS2009-101
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: PD-1; VEGFA; CTLA4; tri-specific antibody; advanced solid tumors; Phase I
MeSH Terms: interventions — Pemetrexed; Carboplatin; Paclitaxel; Etoposide; 130-nm albumin-bound paclitaxel; Oxaliplatin; Capecitabine; Docetaxel; Leucovorin; Fluorouracil; Irinotecan; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Participants will be administered escalating doses of CS2009.
  Interventions: Drug: CS2009
- Dose Expansion (Experimental): Participants will be administered the recommended dose(s) of CS2009 with or without chemotherapy according to dose-escalation data.
  Interventions: Drug: CS2009; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel; Drug: Etoposide; Drug: Nab-paclitaxel; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Docetaxel; Drug: Leucovorin; Drug: 5-FU; Drug: Irinotecan; Drug: Cisplatin

INTERVENTIONS:
Drug: CS2009 — CS2009 will be administered via intravenous (IV) infusion on Day 1 of repeated 21-day cycles (Q3W).
  Arms: Dose Escalation
Drug: CS2009 — CS2009 will be administered via intravenous (IV) infusion on Day 1 of repeated 14/21-day cycles (Q2W/Q3W).
  Arms: Dose Expansion
Drug: Pemetrexed — IV infusion
  Arms: Dose Expansion
Drug: Carboplatin — IV infusion
  Arms: Dose Expansion
Drug: Paclitaxel — IV infusion
  Arms: Dose Expansion
Drug: Etoposide — IV infusion
  Arms: Dose Expansion
Drug: Nab-paclitaxel — IV infusion
  Arms: Dose Expansion
Drug: Oxaliplatin — IV infusion
  Arms: Dose Expansion
Drug: Capecitabine — oral tablets
  Arms: Dose Expansion
Drug: Docetaxel — IV infusion
  Arms: Dose Expansion
Drug: Leucovorin — IV infusion
  Arms: Dose Expansion
Drug: 5-FU — IV infusion
  Arms: Dose Expansion
Drug: Irinotecan — IV infusion
  Arms: Dose Expansion
Drug: Cisplatin — IV infusion
  Arms: Dose Expansion

SUMMARY:
This is a first-in-human (FIH), open-label, and multi-center Phase I/II study designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-tumor activity of CS2009 as Monotherapy and Combination Therapy in Participants with Advanced Solid Tumors. The study is comprised of a Phase I dose escalation and Phase II dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Age ≥ 18 years on the day of signing informed consent.

Phase I:

* Pathologically or cytologically confirmed, unresectable advanced solid tumors, including but not limited to non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), renal cell carcinoma (RCC), hepatocellular carcinoma (HCC), gastric cancer (GC), ovarian cancer (OC), cervical cancer (CC), etc.
* Failure of established standard of care for advanced disease, or no available standard of care.

Phase II:

* Pathologically or cytologically confirmed unresectable advanced solid tumors, including non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), etc.
* Participants with at least one measurable lesion as defined per RECIST v1.1 solid tumor.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function.
* Fertile male participants and female participants of childbearing potential must be willing to use an effective method of birth control from providing signed consent and for 180 days after the last investigational product administration.
* Female participants of childbearing potential must have a negative pregnancy test ≤ 7 days prior to the first dose of the investigational product.

Exclusion Criteria:

* History of a second malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured.
* Known primary central nervous system (CNS) tumor or solid tumor CNS metastasis that is either symptomatic, untreated, or requires therapy.
* Presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage within 4 weeks prior to the first dose of investigational product.
* Receipt of systemic corticosteroid treatment or any other form of immune suppressing treatment within 7 days prior to the first dose of investigational product.
* Active or prior history of definite inflammatory bowel disease.
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, or presence of active or suspected ILD/pneumonitis.
* Active infections requiring systemic therapy within 2 weeks prior to the first dose of investigational product.
* Positive for human immunodeficiency virus (HIV) or presence of acquired immune deficiency syndrome (AIDS).
* Active Hepatitis B or C infection.
* Active pulmonary tuberculosis (TB).
* Major surgery, chemotherapy, definitive radiotherapy, target therapy, immunotherapy, or other anti-cancer therapy within 21 days prior to the first dose of investigational product.
* Palliative radiotherapy within 14 days prior to the first dose of investigational product, or receipt of radioactive drug within 56 days prior to the first dose of investigational product.
* Administration of live vaccine within 28 days prior to the first dose of investigational product.
* History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* Receipt of antitumor Chinese herbal preparations or Chinese patent medicine within 7 days prior to the first dose of investigational product.
* Receipt of any other investigational drugs within 21 days prior to the first dose in this trial.
* History of hypersensitivity or idiosyncrasy to the excipients of the study drug or any monoclonal antibody.
* Any toxic effects of prior therapy or surgical procedures unresolved to baseline severity or NCI-CTCAE Version 5.0 Grade ≤ 1.
* Active alcohol or drug abuse.
* Female participants who are pregnant or breastfeeding.
* Other acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or investigational product administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
[Dose Escalation] Maximum tolerated dose (MTD) of CS2009 | Cycle 1 (Up to 21 Days)
  Participants will receive CS2009 via intravenous (IV) infusion on Day 1 of repeated 21-day cycles (Q3W). The MTD will be determined, if any, by the number of participants who experience a dose limiting toxicity (DLT).
[Dose Escalation] Tentative recommended Phase II dose (RP2D) of CS2009 | Cycle 1 (Up to 21 Days)
  The selection of tentative RP2D will be based on consideration of overall safety information together with available pharmacokinetic, pharmacodynamic, and efficacy data. The tentative RP2D may be the MTD or a lower dose within the tolerable dose range.
[Dose Escalation] Number of participants with adverse events (AEs) | Up to approximately 2 years
[Dose Expansion] Objective response rate (ORR) evaluated by investigators per RECIST v1.1 | Up to approximately 2 years

SECONDARY OUTCOMES:
[Dose Escalation & Expansion] Area under the curve (AUC) of CS2009 | Up to approximately 2 years
[Dose Escalation & Expansion] Maximum concentration (Cmax) of CS2009 | Up to approximately 2 years
[Dose Escalation & Expansion] Elimination half-life (t1/2) of CS2009 | Up to approximately 2 years
[Dose Escalation & Expansion] Minimum concentration (Cmin) of CS2009 | Up to approximately 2 years
[Dose Escalation & Expansion] Number of participants with anti-CS2009 antibodies | Up to approximately 2 years
[Dose Escalation] Objective response rate (ORR) evaluated by investigators per RECIST v1.1 | Up to approximately 2 years
[Dose Expansion] Number of participants with adverse events (AEs) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (30):
- Australia (8):
  - Alfred Hospital (Alfred Health), Melbourne
  - Austin Hospital (Austin Health), Melbourne
  - Monash Medical Centre (Monash Health), Melbourne
  - Peter Maccallum Cancer Centre Research, Melbourne
  - Icon Cancer Centre South Brisbane, South Brisbane
  - Blacktown Hospital, Sydney
  - Macquarie University Hospital, Sydney
  - Scientia Clinical Research Ltd, Sydney
- China (22):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Hospital, Hefei
  - Central Hospital Affiliated to Shandong First Medical University, Jinan
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Xuzhou Central Hospital, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No